CLINICAL TRIAL: NCT00002241
Title: A Multicenter, Open-Label, 24-Week Pilot Study to Evaluate the Safety and Efficacy of Indinavir Sulfate 800 Mg b.i.d. in Combination With Ritonavir 100 Mg/d4T/3TC b.i.d. in HIV-Infected Individuals
Brief Title: Safety and Effectiveness of an Anti-HIV Drug Combination Taken Twice Daily
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246T; 094-00; CRX463
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-07

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Ritonavir; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to see whether taking indinavir (IDV) plus ritonavir (RTV) plus stavudine (d4T) plus lamivudine (3TC) 2 times each day is safe and can lower the level of HIV in the blood.

DETAILED DESCRIPTION:
Patients take IDV plus RTV plus d4T plus 3TC twice daily for 24 weeks. Every 4 weeks, patients have physical exams and laboratory tests of blood and urine, and CD4 cell counts and plasma viral RNA are measured. At Week 24, the proportion of patients with plasma viral RNA below 400 copies/ml is determined to identify any clinically meaningful antiretroviral activity for the drug regimen. An observed response proportion of 80% or higher will be considered clinically meaningful.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a CD4 cell count of 75 cells/mm3 or more and a viral load of 5,000 copies/ml or more.
* Are age 16 or older (consent of a parent or guardian required if under 18).
* Agree to practice abstinence or use barrier methods of birth control (such as condoms).
* Are willing to stop taking all anti-HIV drugs except study drugs. (Patients may be able to continue taking drugs for other infections.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have cancer, lung disease, severe hepatitis, or active AIDS-related infections. (Certain AIDS-related infections such as Kaposi's sarcoma may be allowed).
* Have ever taken 3TC, abacavir (ABC), or a protease inhibitor (such as IDV or RTV).
* Have changed their medications in the last 2 weeks.
* Are allergic to IDV, RTV, d4T, or 3TC.
* Have used certain medications (see the technical summary for more detail).
* Are pregnant or breast-feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Apogee Med Group, San Diego, California
  - Univ of California at San Francisco Gen Hosp, San Francisco, California
  - HIV Institute / Davies Med Ctr, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - Univ of Miami School of Medicine, Miami, Florida
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - CRI New England, Brookline, Massachusetts
  - SUNY Health Sciences Ctr, Brooklyn, New York
  - Chelsea Village Med Ctr, New York, New York
  - Liberty Med Group, New York, New York
  - St Lukes / Roosevelt Hosp / HIV Center, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Montefiore Med Ctr, The Bronx, New York
  - Mark Watkins, Philadelphia, Pennsylvania
  - Univ of Texas / Thomas Street Clinic, Houston, Texas